CLINICAL TRIAL: NCT01179022
Title: Incidence of Bacteremia Following Argon Plasma Coagulation in Patients With Endobronchial Lesions
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10-137-10.CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Bacteremia
Keywords: Bacteremia; Argon Plasma Coagulation; Endobronchial Lesions
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Incidence of Bacteremia Following Argon Plasma Coagulation in Patients with Endobronchial Lesions

DETAILED DESCRIPTION:
Bacteremia is a well-recognized invasive medical condition. In most cases, it is a transient phenomenon without clinical consequences. In certain patients, such as those with structural cardiac abnormalities, it may lead to the development of infectious endocarditis. According to an American Heart Association statement, routine endocarditis prophylaxis is indicated prior to invasive procedures with relatively high bacteremia rates, such as dental care,certain types of catheterization and rigid bronchoscopy [1].Fibreoptic bronchoscopy, with or without biopsy is not included in this list due to a very low bacteremia rate [1].This even applies to particularly high risk patients with prosthetic valve or previous endocarditis. Yigla et al. assessed the incidence of bacteremia following bronchoscopy and found 6.5% of bacteremia rate. (2) Recently, Steinfort et al. assessed the bacteremia rate following endobronchial ultrasound and found 7% of bacteremia rate following the procedure. All bacterial isolates were typical oropharyngeal commensal organisms. The transbronchial needle aspiration washing culture was positive in 35% of the patients. However, none of the bacteremic patients had clinical features suggestive of infection and no complications were seen among the cohort. (3) No data are available, however about the bacteremic rate following interventional bronchoscopy for endobronchial obstruction and advance lung carcinoma. In these cases, palliative setting of alleviating central airway obstruction, laser resection, electrocautery, argon plasma coagulation and stenting are techniques that can provide immediate relief.

Argon plasma coagulation (APC) is uses ionize argon gas jet flow to conduct electrons allowing a noncontact mode of treatment (lightning effect). (4, 5) APC has been popular in gastrointestinal endoscopy for superficial coagulation of large mucosal surfaces. The argon gas quite flexibly flows around bends and corners. Coagulated tissue has a higher resistance that automatically drives the argon gas flow away to nearby untreated tissue. An immediate effect really can be seen during electrocautery treatment, which corresponds well with the histological effect of coagulative necrosis.

We therefore conduct a prospective study to assess the bacteremic rate following APC in patients with endobronchial involvement.

ELIGIBILITY:
Inclusion Criteria:

* All patients that undergo bronchoscopy with the use of APC

Exclusion Criteria:

* All patients under 18 years old All Patients with evidence of current respiratory infection or febrile illnesses and those that will receive antibiotic therapy within a week prior to the bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients that undergo bronchoscopy with the use of APC
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The bacteremic rate following APC in patients with endobronchial involvment. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: DAVID SHITRIT, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir MC, Kfar Saba, Israel, Israel

REFERENCES:
- [Derived] Matveychuk A, Guber A, Talker O, Shitrit D. Incidence of bacteremia following bronchoscopy with argon plasma coagulation: a prospective study. Lung. 2014 Aug;192(4):615-8. doi: 10.1007/s00408-014-9583-8. Epub 2014 Apr 27. PMID 24770443